CLINICAL TRIAL: NCT04174482
Title: Pilot Study of Morphological and Functional Evaluation of Adult Flat Foot by Weight Bearing CT and Gait Analysis Before and After Corrective Surgery
Brief Title: Morphological and Functional Evaluation of Adult Flat Foot Before and After Corrective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBCT-PIEDE PIATTO
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2019-11

CONDITIONS: Flat Feet
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flat foot patients (Experimental): 20 patients recruited consecutively and candidates for surgery to correct the adult flat foot according to the Grice technique.
  Interventions: Procedure: morphological and functional evaluation of adult flat foot

INTERVENTIONS:
Procedure: morphological and functional evaluation of adult flat foot — Evaluations are realized by weight bearing computed tomography and by Gait analysis in the pre-operative phase and at a 6-months follow-up from the surgery with Grice technique

SUMMARY:
Morphological weight bearing computed tomography parameters and gait analysis can implement the evaluation of the flat foot. Weight bearing CT is useful to verify the severity of the 3D deformities typical of flat foot, while kinematic and kinetic variables of gait is able to quantify the functional improvements of the foot after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with idiopathic flat foot with indication for corrective surgical treatment according to Grice (arthrodesis of the subtalar joint)
* age between 18 and 65 years
* BMI less than 40
* signature of informed consent.

Exclusion Criteria:

* patients with severe alterations or other pathologies affecting the foot and lower limb
* severe vascular and neurological systemic diseases
* systemic diseases that can compromise bone consolidation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Weight bearing computed tomography parameter | change from baseline at 6-months
  calcaneal pitch angle (degree)
Gait Analysis parameter | change from baseline at 6-months
  medial longitudinal arch

SECONDARY OUTCOMES:
Pain clinical examination parameter | pre-operative phase and at a 6-months follow-up from the intervention
  visual analogue scale of the foot
Posture clinical examination parameter | pre-operative phase and at a 6-months follow-up from the intervention
  Foot Posture Index
Function clinical examination parameter | pre-operative phase and at a 6-months follow-up from the intervention
  Foot function Index

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Burssens A, Peeters J, Buedts K, Victor J, Vandeputte G. Measuring hindfoot alignment in weight bearing CT: A novel clinical relevant measurement method. Foot Ankle Surg. 2016 Dec;22(4):233-238. doi: 10.1016/j.fas.2015.10.002. Epub 2015 Oct 30. PMID 27810020
- [Result] Buldt AK, Levinger P, Murley GS, Menz HB, Nester CJ, Landorf KB. Foot posture is associated with kinematics of the foot during gait: A comparison of normal, planus and cavus feet. Gait Posture. 2015 Jun;42(1):42-8. doi: 10.1016/j.gaitpost.2015.03.004. Epub 2015 Mar 12. PMID 25819716
- [Result] Leardini A, Benedetti MG, Berti L, Bettinelli D, Nativo R, Giannini S. Rear-foot, mid-foot and fore-foot motion during the stance phase of gait. Gait Posture. 2007 Mar;25(3):453-62. doi: 10.1016/j.gaitpost.2006.05.017. Epub 2006 Sep 11. PMID 16965916

DOCUMENTS (1):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT04174482/Prot_000.pdf